CLINICAL TRIAL: NCT00767585
Title: An Open Label Non-Interventional Evaluation of the Effect of Adjuvant Hormonal Treatment of Postmenopausal Women Wih Early Breast Cancer With Aromatase Inhibitors on Bone Mineral Density and Bone Fracture Rate in Daily Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Meta Jeras, Mr Ph, Regulatory and Medical Affairs Manager, AstraZeneca UK Limited, Branch Office in Slovenia
Other Study IDs: NIS-OSI-DUM-2008/1
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: breast cancer; aromatase inhibitors; bone mineral density; osteoporosis
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- A:: 70 women with hormone-dependent or hormone-independent early breast cancer that have completed their chemo- and/or radiotherapy just recently (up to 6 months after completion of therapy)
- B: 70 women with hormone-independent early breast cancer, 24-36 months after completion of chemo- and/or radiotherapy
- C: 70 women with hormone-independent early breast cancer, 54-66 months after completion of chemo- and/or radiotherapy
- D: 70 women with hormone-dependent early breast cancer, 24-36 months after initiation of tamoxifen therapy
- E: 70 women with hormone-dependent early breast cancer, 24-36 months after initiation of aromatase inhibitors therapy
- F: 70 women with hormone-dependent early breast cancer, 54-66 months after initiation of tamoxifen therapy
- G: 70 women with hormone-dependent early breast cancer, 54-66 months after initiation of aromatase inhibitors therapy
- H: 70 women with hormone-dependent early breast cancer, 24-36 months after initiation of aromatase inhibitors therapy following 24-36 months of initial tamoxifen therapy

SUMMARY:
The aim of this study is to determine the effect of aromatase inhibitors therapy on bone mineral density and compare it to the effects of tamoxifen and no hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 55-65 years, diagnosed with invasive early breast cancer: - Surgery, chemo- and/or radiotherapy concluded less than 6 months ago
* Women with hormone-independent breast cancer: - Surgery, chemo- and/or radiotherapy concluded before 24-36 months or 54-66 months
* Women with hormone-dependent breast cancer:- Adjuvant therapy with tamoxifen initiated before 24-36 and 54-66 months or - Adjuvant therapy with aromatase inhibitor initiated before 24-36 and 54-66 months or - Switch from tamoxifen to aromatase inhibitor initiated before 24-36 months

Exclusion Criteria:

* Women receiving active treatment for osteoporosis
* Women with any evidence of breast cancer recurrence

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Institute of Oncology
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2008-08; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine the effect of aromatase inhibitors therapy on bone mineral density as measured by DEXA scan and compare it to the effects of tamoxifen and no hormonal therapy. | once

SECONDARY OUTCOMES:
To determine the bone fracture rate in women on aromatase inhibitors therapy and compare it to fracture rates observed in the tamoxifen and the hormone-independent group. | once

CONTACTS AND LOCATIONS:
Overall Officials: Simona Borstnar, MD, PhD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Research Site, Ljubljana, Slovenia